CLINICAL TRIAL: NCT01210911
Title: A Phase II, Randomized, Placebo Controlled Study to Evaluate the Efficacy of the Combination of Gemcitabine, Erlotinib and Metformin in Patients With Locally Advanced and Metastatic Pancreatic Cancer
Brief Title: Metformin Combined With Chemotherapy for Pancreatic Cancer
Acronym: GEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.W. Wilmink, Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMCmedonc10/003
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Locally Advanced Pancreatic Cancer; Metastatic Pancreatic Cancer
Keywords: pancreatic cancer; metformin; MAPK pathway; PI3K/Akt pathway; gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Erlotinib Hydrochloride; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine, erlotinib and metformin (Experimental): Gemcitabine at a dose of 1000 mg/m2 (iv, 30 minutes) will be given weekly, for 3 weeks, followed by one week without gemcitabine. Erlotinib will be administered at a daily dose of 100 mg at least one hour before or 2 hours after the ingestion of food. Metformin will be administered at a dose of 500 mg twice daily. If well tolerated the dose will be increased to 1000 mg twice daily in the second week.
  Interventions: Drug: gemcitabine; Drug: erlotinib; Drug: metformin
- Gemcitabine, erlotinib and placebo (Placebo Comparator): Gemcitabine at a dose of 1000 mg/m2 (iv, 30 minutes) will be given weekly, for 3 weeks, followed by one week without gemcitabine. Erlotinib will be administered at a daily dose of 100 mg at least one hour before or 2 hours after the ingestion of food. PLacebo will be administered at a dose of 500 mg twice daily. If well tolerated the dose will be increased to 1000 mg twice daily in the second week.
  Interventions: Drug: gemcitabine; Drug: erlotinib; Drug: placebo

INTERVENTIONS:
Drug: gemcitabine — Gemcitabine at a dose of 1000 mg/m2 (iv, 30 minutes) will be given weekly, for 3 weeks, followed by one week without gemcitabine
  Other Names: gemzar
Drug: erlotinib — Erlotinib will be administered at a daily dose of 100 mg at least one hour before or 2 hours after the ingestion of food
  Other Names: Tarceva
Drug: metformin — Metformin will be administered at a dose of 500 mg twice daily for the first week. If tolerated well, the dose will be increased up to 1000 mg twice daily in the second week.
  Other Names: Glucophage
  Arms: Gemcitabine, erlotinib and metformin
Drug: placebo — Placebo will be administered at a dose of 500 mg twice daily for the first week. If tolerated well, the dose will be increased up to 1000 mg twice daily in the second week.
  Arms: Gemcitabine, erlotinib and placebo

SUMMARY:
Pancreatic cancer patients have one of the worst prognoses among all cancer types with a 5 year survival rate of less than 5%. Despite significant changes during the last decade in our molecular knowledge on this disease, the prognosis and management of pancreatic cancer have remained unchanged. With the advances in molecular biology, newer biologic agents such as erlotinib, are adding some benefit to the conventional cytotoxic agents. There is a growing body of literature suggesting that type 2 diabetes mellitus (DM) may be associated with the development of pancreatic cancer, but this association is complex. Because various DM medications can affect directly the key factors mediating the association between DM and pancreatic cancer, understanding the effect of anti-diabetic therapies on pancreatic cancer is a critical step in fully characterizing the role of type 2 DM in the development of pancreatic cancer. Indeed, two epidemiologic studies have found that diabetic patients treated with metformin were less likely to develop cancer, but those treated with insulin were more likely to die of various kinds cancer. Not only does metformin ameliorate hyperglycemia and hyperinsulinemia, both of which are associated with the adverse impact of DM on cancer, metformin also has direct metabolic effects through activation of adenosine monophosphate-activated protein kinase (AMPK). AMPK regulates many metabolic enzymes and also inhibits the mammalian target of rapamycin (mTOR) pathway via phosphorylation and stabilization of the tumor suppressor gene TSC2. But there is an intensive cross-talk between various pathways. Inhibition of the phosphoinositide 3-kinase (PI3K)/Akt pathway, of which mTOR is one of the effector proteins, for instance may result in escape via the mitogen-activated protein kinase (MAPK) pathway and vice verse. Indeed, epidermal growth factor receptor (EGFR) activation leads to activation of the MAPK pathway and the PI3K pathway. Thus, since it is clear that blocking one pathway will not always be sufficient to produce a response in the presence of other activated pathways, the best change of success will be realized when using a combination of agents that inhibit separate pathways known to be critical to the survival of the tumour. In line with these observations, combining a small molecule against the EGFR and inhibition of the PI3K pathway by metformin might account for potential candidates of the above combinatorial approach. Therefore, in this study, the investigators want to determine the activity and safety of concurrent interruption of the MAPK and PI3K pathways by the EGFR tyrosine kinase inhibitor erlotinib and metformin, combined with gemcitabine in patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
In this phase II randomized, placebo controlled study, patients with locally advanced or metastatic pancreatic cancer will be randomized to treatment with gemcitabine, erlotinib and metformin, or gemcitabine, erlotinib and placebo.

Gemcitabine at a dose of 1000 mg/m2 (iv, 30 minutes) will be given weekly, for 3 weeks, followed by one week without treatment. Erlotinib will be administered at a daily dose of 100 mg at least one hour before or 2 hours after the ingestion of food. Metformin/ placebo will be administered at a dose of 500 mg twice daily. If well tolerated the dose will be increased to 1000 mg twice daily in the second week.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed content obtained prior to treatment
* Cytological or histological confirmed carcinoma of the pancreas
* Metastatic cancer
* Measurable lesion according to RECIST criteria
* ECOG/ WHO performance 0-2
* Age > 18 years
* Adequate renal function (creatinine < 150 µmol/L and/ or a creatinine clearance > 60 ml/ L)
* Adequate liver function (bilirubin < 1.5 times upper limit of normal, ALAT or ASAT < 5.0 times upper limit of normal in case of liver metastases and < 2.5 the upper limit of normal in absence of liver metastases).
* Adequate bone marrow function (WBC > 3.0 x 10 9/L, platelets > 100 x 10 9/L)
* Mentally, physically, and geographically able to undergo treatment and follow up

Exclusion Criteria:

* Clinical or radiological evidence of CNS metastases
* Pregnancy (positive serum pregnancy test) and lactation
* Serious concomitant systemic disorder that would compromise the safety of the patient, at the discretion of the investigator
* Patients who have any severe and/or uncontrolled medical conditions:

  * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤ 6 months prior to randomization, serious uncontrolled cardiac arrhythmia
  * uncontrolled diabetes as defined by fasting serum glucose >2X ULN.
  * active or uncontrolled severe infection.
  * cirrhosis, chronic active hepatitis or chronic persistent hepatitis
  * severely impaired lung function
* Previous treatment with erlotinib
* Previous treatment with gemcitabine for metastatic disease
* Previous treatment with gemcitabine combined with radiotherapy for locally advanced pancreatic cancer within 6 months prior to study entry
* Patients with a known hypersensitivity to metformin
* Use of metformin in the previous 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-08; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Survival after 6 months | 6 months after completion of the study

SECONDARY OUTCOMES:
Progression free survival | 6 months after the completion of the study
Objective response rate | expected treatment duration 2- 6 months
toxicity profile | during study and 4 weeks after stop study medication

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke Wilmink, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Kordes S, Pollak MN, Zwinderman AH, Mathot RA, Weterman MJ, Beeker A, Punt CJ, Richel DJ, Wilmink JW. Metformin in patients with advanced pancreatic cancer: a double-blind, randomised, placebo-controlled phase 2 trial. Lancet Oncol. 2015 Jul;16(7):839-47. doi: 10.1016/S1470-2045(15)00027-3. Epub 2015 Jun 8. PMID 26067687